CLINICAL TRIAL: NCT06167720
Title: Suicide Risk Prediction in Cancer Patients: a Retrospective Cohort Study
Brief Title: Suicide Risk Prediction in Cancer Patients
Status: Completed | Type: Observational
Sponsor: Fang Tang (Other)
Responsible Party: Sponsor-Investigator, Fang Tang, Doctor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2023(139)
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Cancer
Keywords: Cancer patients; Suicide risk; Prediction model; Meteorological factors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer patients cohort in SEER database: A retrospective cohort of cancer patients based on the Surveillance, Epidemiology, and End Results (SEER) program database was used to assess the association of socioeconomic factors, clinical characteristics and meteorological factors with cancer patients' suicide, and to establish prediction model with multiple predictors for cancer patient
- Cancer patients cohort in SMCHBDP: Retrospective cohort conducted from Shandong Multi-Center Healthcare Big Data Platform (SMCHBDP) was used to verify the predictive ability and generalization ability of the prediction model.

SUMMARY:
Previous studies have found that the suicide risk of cancer patients is influenced by socioeconomic factors, clinical characteristics, and environmental factors. But prediction model with multiple predictors for suicide risk in cancer patients is limited.

The aim of this study is to assess the association of socioeconomic factors, clinical characteristics and meteorological factors with cancer patients' suicide, based on retrospective cohorts, and to establish a suicide risk prediction model with multiple predictors for cancer patients.

DETAILED DESCRIPTION:
Cancer is a serious public health concern, with almost 10 million people dying from cancer in 2020. Previous studies have reported that cancer patients are more likely to die by suicide than the general public, especially in the six months to one year following cancer diagnosis. Since suicide is a result of the interaction of various factors such as socioeconomic factors, clinical characteristics, and environmental factors, it is necessary to construct a multivariate prediction model to predict the suicide risk in cancer patients.

A retrospective cohort of cancer patients based on the Surveillance, Epidemiology, and End Results (SEER) program database was used to assess the association of socioeconomic factors, clinical characteristics and meteorological factors with cancer patients' suicide, and to establish prediction model with multiple predictors for cancer patients. Another retrospective cohort conducted from Shandong Multi-Center Healthcare Big Data Platform (SMCHBDP) was used to verify the predictive ability and generalization ability of the prediction model.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients in SEER database and SMCHBDP

Exclusion Criteria:

1. No certain cause of death
2. Missing area code
3. Lost to follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cancer patients in the Surveillance, Epidemiology, and End Results (SEER) program database and Shandong Multi-Center Healthcare Big Data Platform (SMCHBDP).
Sampling Method: Non-Probability Sample
Enrollment: 176000 (Actual)
Dates: Start 1979-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality attributed to suicide or self-inflicted injury | 1979-2021
  The main outcome was mortality attributed to suicide or self-inflicted injury after cancer diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Tang, Doctor, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China